CLINICAL TRIAL: NCT04475705
Title: The Effects of Propofol Based Intravenous vs Sevoflurane Inhalation Anaesthesia on Inflammation and Circulating Tumor Cells in Paediatric Tumor Surgery - a Pilot Study
Brief Title: Propofol vs Sevo for Paediatric Tumor Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hong Kong Children's Hospital (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKCH-REC-2020-013
Record Dates: First submitted 2020-07-07; First posted 2020-07-17 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Solid Tumor; Carcinoma; Malignancy; Cancer
Keywords: propofol; sevoflurane; cancer surgery; circulating tumor cells; paediatric
MeSH Terms: conditions — Carcinoma; Neoplasms; Neoplastic Cells, Circulating | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: single blind controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sevoflurane group (Active Comparator): patients in this group will receive inhalation anaesthesia with sevoflurane at Minimal Alveolar Concentration 0.7-1.3 as the main anaesthetic to achieve Bispectral Index 40-60. Other anaesthetic management will be standardised.
  Interventions: Drug: sevoflurane
- propofol group (Active Comparator): patients in this group will receive intravenous propofol using Target Controlled Infusion 'Paedfusor' model 2-5 as the main anaesthetic to achieve Bispectral Index 40-60. Other anaesthetic management will be standardised.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — intravenous propofol using Target Controlled Infusion 'Paedfusor' model 2-5 as the main anaesthetic to achieve Bispectral Index 40-60
  Other Names: Diprivan
  Arms: propofol group
Drug: sevoflurane — sevoflurane at Minimal Alveolar Concentration 0.7-1.3 as the main anaesthetic to achieve Bispectral Index 40-60.
  Other Names: ultane, sevorane
  Arms: Sevoflurane group

SUMMARY:
Background:

Retrospective studies and meta-analyses have shown a reduction in 5-year survival following inhalational based compared to propofol based total intravenous (TIVA) anaesthesia for cancer surgery. To date there have been no prospective trials published which evaluate the effect of anaesthetic technique on circulating tumour cells (CTC), oxidative stress, and recurrence rate following cancer surgery. Children with cancer often require surgery for tumour excision as well as for other diagnostic and therapeutic procedures. To date there has been no prospective randomized controlled trial evaluating the optimal anaesthetic technique for surgery on children with cancer.

Aim:

This is a pilot study in paediatric patients who require surgery for tumour excision. The aim is to investigate the effect of sevoflurane inhalational versus propofol intravenous anaesthesia on expression of hypoxia-inducible factor 1 (HIF-1), circulating tumour cells, DNA damage and biomarkers of immunity and inflammation in patients before and after tumour surgery. The patients will be followed up for up to 5 years for tumour recurrence after surgery.

Method:

This will be a single-blinded randomized controlled trial. One hundred children undergoing tumour excision surgery at the Hong Kong Children's Hospital will be recruited and randomized to receive TIVA or inhalational anaesthesia. Baseline, intraoperative and postoperative blood will be taken for tests of immunity and inflammatory markers, DNA damage and circulating tumour cells. Patients would be followed up to 3 years for tumour recurrence and survival.

DETAILED DESCRIPTION:
Surgical resection is the main modality of treatment for many solid tumors. Despite successful tumor resection, some patients develop local recurrence or metastasis, causing morbidities and mortality. In recent years, there is growing interest in the pathophysiology of recurrence or metastasis. It is believed that the recurrence is caused by the liberation of circulating tumor cells during surgical manipulation of the tumors and the vascular invasive properties of the tumor cells. Perioperative events, such as surgical stress and anaesthesia may have immunomodulating effects, causing growth or inhibition of circulating tumor cells, which affect disease relapse. There is growing evidence that propofol is anti-inflammatory while sevoflurane is pro-inflammatory and their potential roles in cancer recurrence attract researchers' attention. In adults, there is increasing number of researches showing that propofol may improve patient outcomes in terms of disease survival, when compared to sevoflurane. However, such evidence in paediatric population is lacking. This study aims to compare the effects of propofol based intravenous anaesthesia with inhalation anaesthesia with sevoflurane on perioperative biomarkers of inflammation, circulating tumor cells and disease free survival in 3 years.

100 patients will be recruited for this single blinded randomised controlled trial. They will receive general anaesthesia in Hong Kong Children's Hospital for their primary tumor excision surgery. 50 patients will be randomised to sevoflurane group and 50 patients will be randomised to propofol group. They will receive standardised anaesthetic management in terms of death or anaesthesia, pain management, fluid or thermoregulation management. Sevoflurane group subjects will receive inhalational sevoflurane as main anaesthetic, while propofol group subjects will receive intravenous propofol. These patients will have 4 blood tests collected for analysis for biomarkers of inflammation, DNA damage, oxidative stress and circulating tumor cells.

* baseline: once patients have intravenous access established
* intraoperative: when the tumor is deemed resected by surgeons
* immediately postop: after wound closure
* 24 hours postop Early postoperative period follow up will look for wound recovery, sepsis, and time to start chemotherapy and need for second look operation for wound complication.

Patients will also followed up for 3 years for tumor recurrence and disease survival.

ELIGIBILITY:
Inclusion Criteria:

* patients coming for elective primary solid tumor resection for curative intent in Hong Kong Children's Hospital
* AND patients > 5kg
* AND patients within age limit

Exclusion Criteria:

* Autoimmune / Chronic inflammatory diseases e.g. Systemic Lupus Erythematosus (SLE), Rheumatoid Arthritis (RA) etc.
* Current Steroid therapy
* Surgery for tumour removal in the past year
* Allergy to Propofol
* intraoperative use of nitrous oxide
* Patient susceptible to Malignant Hyperthermia
* Patients / parents / legal guardians showing preference in anaesthetic techniques during recruitment process

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
difference in Hypoxia Inducible Factor-1 gene expression | intraoperative to postoperative 24 hours
  pg/mL

SECONDARY OUTCOMES:
difference in levels of Interleukin-6 | intraoperative to postoperative 24 hours
  pg/mL
difference in levels of Tumor Necrosis Factor-alpha | intraoperative to postoperative 24 hours
  pg/mL
difference in levels of high sensitivity C reaction protein | intraoperative to postoperative 24 hours
  mg/L
difference in levels of DNA damage (Comet Assay) | intraoperative to postoperative 24 hours
  %T (percent tail)
difference in levels of Glutathione Peroxidase | intraoperative to postoperative 24 hours
  μg/mL
difference in levels of Superoxide dismutase | intraoperative to postoperative 24 hours
  units/ml
difference in levels of urinary 8-oxo-7,8-dihydro-2'-deoxyguanosine (8-oxodG) | intraoperative to postoperative 24 hours
  ng/mL
difference in levels of 8-oxo-7,8-dihydroguanosine (8-oxoGuo) | intraoperative to postoperative 24 hours
  ng/mL
difference in the quantity of circulating tumor cells (CTC) | intraoperative to postoperative 24 hours
  cells/100 µL
cancer free survival at 1 and 3 years | intraoperative to postoperative 24 hours
  percent

CONTACTS AND LOCATIONS:
Overall Officials: Sau Man Lee, MBBS, Principal Investigator — Hong Kong Children's Hospital
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Divatia JV, Ambulkar R. Anesthesia and cancer recurrence: What is the evidence? J Anaesthesiol Clin Pharmacol. 2014 Apr;30(2):147-50. doi: 10.4103/0970-9185.129990. No abstract available. PMID 24803747
- [Background] Heaney A, Buggy DJ. Can anaesthetic and analgesic techniques affect cancer recurrence or metastasis? Br J Anaesth. 2012 Dec;109 Suppl 1:i17-i28. doi: 10.1093/bja/aes421. PMID 23242747
- [Background] Vinay DS, Ryan EP, Pawelec G, Talib WH, Stagg J, Elkord E, Lichtor T, Decker WK, Whelan RL, Kumara HMCS, Signori E, Honoki K, Georgakilas AG, Amin A, Helferich WG, Boosani CS, Guha G, Ciriolo MR, Chen S, Mohammed SI, Azmi AS, Keith WN, Bilsland A, Bhakta D, Halicka D, Fujii H, Aquilano K, Ashraf SS, Nowsheen S, Yang X, Choi BK, Kwon BS. Immune evasion in cancer: Mechanistic basis and therapeutic strategies. Semin Cancer Biol. 2015 Dec;35 Suppl:S185-S198. doi: 10.1016/j.semcancer.2015.03.004. Epub 2015 Mar 25. PMID 25818339
- [Background] Demicheli R, Retsky MW, Hrushesky WJ, Baum M, Gukas ID. The effects of surgery on tumor growth: a century of investigations. Ann Oncol. 2008 Nov;19(11):1821-8. doi: 10.1093/annonc/mdn386. Epub 2008 Jun 10. PMID 18550576
- [Background] Tavare AN, Perry NJ, Benzonana LL, Takata M, Ma D. Cancer recurrence after surgery: direct and indirect effects of anesthetic agents. Int J Cancer. 2012 Mar 15;130(6):1237-50. doi: 10.1002/ijc.26448. Epub 2011 Nov 9. PMID 21935924
- [Background] Benzonana LL, Perry NJ, Watts HR, Yang B, Perry IA, Coombes C, Takata M, Ma D. Isoflurane, a commonly used volatile anesthetic, enhances renal cancer growth and malignant potential via the hypoxia-inducible factor cellular signaling pathway in vitro. Anesthesiology. 2013 Sep;119(3):593-605. doi: 10.1097/ALN.0b013e31829e47fd. PMID 23774231
- [Background] Kushida A, Inada T, Shingu K. Enhancement of antitumor immunity after propofol treatment in mice. Immunopharmacol Immunotoxicol. 2007;29(3-4):477-86. doi: 10.1080/08923970701675085. PMID 18075859
- [Background] Huitink JM, Heimerikxs M, Nieuwland M, Loer SA, Brugman W, Velds A, Sie D, Kerkhoven RM. Volatile anesthetics modulate gene expression in breast and brain tumor cells. Anesth Analg. 2010 Dec;111(6):1411-5. doi: 10.1213/ANE.0b013e3181fa3533. Epub 2010 Oct 1. PMID 20889943
- [Background] Wigmore TJ, Mohammed K, Jhanji S. Long-term Survival for Patients Undergoing Volatile versus IV Anesthesia for Cancer Surgery: A Retrospective Analysis. Anesthesiology. 2016 Jan;124(1):69-79. doi: 10.1097/ALN.0000000000000936. PMID 26556730